CLINICAL TRIAL: NCT01666431
Title: Single-center Investigator Initiated Pilot Study Investigating the Tumor Response of Squamous Cell Carcinoma Lesions in Patients Under Lapatinib Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ10ON03
Record Dates: First submitted 2012-08-08; First posted 2012-08-16 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Lapatinib

ARMS (1):
- Lapatinib (Other)
  Interventions: Drug: Lapatinib

INTERVENTIONS:
Drug: Lapatinib

SUMMARY:
Primary cutaneous squamous cell carcinomas (SCCs) are epithelial carcinomas with a high frequency of EGF-R expression. EGFR is an important regulator of tumour progression and proliferation in several types of cancer. Mechanism of action of Lapatinib in the EGFR and/or HER2 expressing oesophageal squamous cell carcinoma (ESCC) cells is attributed to inhibition of cell proliferation and induction of apoptosis. Based on the data from oesophageal SCCs the investigators hypothesise that EGFR signalling pathway and its interactions play an important role in the SCC pathogenesis and represent a good therapeutic target from these tumours.

Primary Objectives:

To evaluate the tumour response macroscopically in patients with primary cutaneous SCC lesions and in concomitant SCC in situ (AK).

Secondary Objectives:

* To evaluate tolerability of a single dose regimen of systemic lapatinib therapy in patients with SCC as measured by time to first AE or SAE within the study period.
* To investigate the molecular tumour response of squamous cell carcinoma lesions in patients under lapatinib treatment using a set of variables.
* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Diagnosis of histologically confirmed cutaneous SCC stage Tis-T2N0 for which surgical treatment is considered suitable.
* In case of SCC, patients must present with a minimum of two co-existing AK lesions. In case of Keratoacanthoma, one lesion of sufficient size (=1cm) is acceptable.
* All included patients must have both FFPE and frozen material available.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ system function

Exclusion criteria:

* Subjects who have current active hepatic or biliary disease
* Other non-controlled malignancy
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of study treatment.
* Presence of uncontrolled infection
* History of any one or more of the following cardiovascular conditions within the past 6 months:Cardiac angioplasty or stenting;Myocardial infarction;Unstable angina;Coronary artery bypass graft surgery;Symptomatic peripheral vascular disease; Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Prior exposure to the study drug lapatinib
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Macroscopic evaluation of tumour response | 84 days
  The primary efficacy objective is to evaluate the tumour response macroscopically in patients with primary cutaneous SCC lesions and in concomitant SCC in situ (AK) by documenting changes in quantity and two-dimensional measurements (mm).

SECONDARY OUTCOMES:
Evaluation of tolerability | 84 days
  Evaluation of tolerability of a single dose regimen of systemic lapatinib therapy in patients with SCC as measured by time to first AE or SAE within the study period
Molecular evaluation of tumour response | 84 days
  Investigation of molecular tumour response of squamous cell carcinoma lesions in patients under lapatinib treatment using a set of variables

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Dummer, Professor MD, Principal Investigator — University Hospital Zurich, Division of Dermatology
Locations (1):
- University Hospital Zurich, Division of Dermatology, Zurich, Canton of Zurich, Switzerland